CLINICAL TRIAL: NCT03636139
Title: Effects of Transcranial Direct Current Stimulation on the Cognitive Control of Negative Stimuli in Borderline Personality Disorder
Brief Title: Cognitive Control of Negative Stimuli in BPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Freie Universität Berlin (Other)
Responsible Party: Principal Investigator, Lars Schulze, Principal investigator, Freie Universität Berlin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: tDCS_BPD
Record Dates: First submitted 2018-08-10; First posted 2018-08-17 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal stimulation (Experimental): transcranial DC stimulation : anodal
  Interventions: Device: transcranial DC stimulation : anodal
- Sham stimulation (Sham Comparator): transcranial DC stimulation : sham
  Interventions: Device: transcranial DC stimulation : sham

INTERVENTIONS:
Device: transcranial DC stimulation : anodal — anodal stimulation of the right dlPFC (i.e. F4) for 20 minutes
  Arms: Anodal stimulation
Device: transcranial DC stimulation : sham — sham stimulation of the right dlPFC (i.e. F4) for 20 minutes
  Arms: Sham stimulation

SUMMARY:
Borderline personality disorder (BPD) is characterized by impairments in the cognitive control of negative information. These impairments in cognitive control are presumably due to blunted activity of the dorsolateral prefrontal cortex (dlPFC) along with enhanced activations of the limbic system. However, the impact of an excitatory stimulation of the dlPFC still needs to be elucidated. In the present study, we therefore assigned 50 patients with BPD and 50 healthy controls to receive either anodal or sham stimulation of the right dlPFC in a double-blind, randomized, between-subjects design.

ELIGIBILITY:
Inclusion Criteria Borderline Personality Disorder:

* Diagnosis of borderline personality disorder

Exclusion Criteria Borderline Personality Disorder:

* Diagnosis of current or previous bipolar disorder
* Diagnosis of current substance dependency
* Diagnosis of current major depression
* Diagnosis of current or previous neurological disorders (e.g., epilepsy)
* Tattoos or scarred skin on the left shoulder or scalp (i.e. F4)

Inclusion Criteria Control Participants:

* No current or previous diagnosis of a mental disorder

Exclusion Criteria Control Participants:

* More than 2 criteria of borderline personality disorder are met
* Diagnosis of current or previous neurological disorders (e.g., epilepsy)
* Intake of psychotropic medication
* Tattoos or scarred skin on the left shoulder or scalp (i.e. F4)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Response latencies | Response latencies were exclusively measured during the assigned interventions, which lasted approx. 20 minutes. No further time points were assessed.
  Response latencies were measured in the context of a delayed working memory task. In this paradigm, each trial started with a fixation cross (1000 ms), followed by the presentation of six target letters (1500 ms), which participants were asked to memorize. After a variable distracter period (i.e., interference duration of 1000, 2000, or 4000 ms), participants were presented a recognition display (until a response was made) and had to decide whether the presented letter was part of the initial set of letters. In half of the trials, the recognition display contained a previously presented target. The distracter period of the experimental paradigm was manipulated with regard to the factors valence (grey background screen, or neutral, or negative stimuli) and interference duration (1000, 2000, or 4000 ms). Neutral and negative affective stimuli were selected from the International Affective Picture System.

IPD SHARING:
Plan to Share IPD: Undecided